CLINICAL TRIAL: NCT03963193
Title: Phase II Trial of Etoposide Plus Cisplatin Compared With Irinotecan Plus Cisplatin for First-line Treatment of Non-primary Pancreatic Metastatic and/or Unresectable Gastrointestinal Neuroendocrine Tumor G3 Type
Brief Title: Etoposide/Cisplatin Compared With Irinotecan/Cisplatin for Advanced Gastrointestinal Neuroendocrine Tumor G3 Type
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-GI-005
Record Dates: First submitted 2019-05-20; First posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Gastrointestinal Neuroendocrine Tumor
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor | interventions — Etoposide; Cisplatin; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etoposide plus Cisplatin (Experimental): Etoposide 100mg/m^2 ivggt on days 1, 2, 3, Cisplatin 25mg/m^2 ivggt on days 1, 2, 3, repeated every 21 days. When the investigator believes that the participant is not suitable for continued medication or the evaluation is progressive disease (PD) according to the RECIST 1.1 standard, the medication is over.
  Interventions: Drug: Etoposide
- Irinotecan plus Cisplatin (Experimental): Irinotecan 65 mg/m^2 ivggt on days 1, 8, Cisplatin 30 mg/m^2 ivggt on days 1, 8, repeated every 21 days. When the investigator believes that the participant is not suitable for continued medication or the evaluation is progressive disease (PD) according to the RECIST 1.1 standard, the medication is over.
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Etoposide — Etoposide 100mg/m^2 ivggt on days 1, 2, 3, Cisplatin 25mg/m^2 ivggt on days 1, 2, 3, repeated every 21 days.
  Other Names: Cisplatin
  Arms: Etoposide plus Cisplatin
Drug: Irinotecan — Irinotecan 65 mg/m^2 ivggt on days 1, 8, Cisplatin 30 mg/m^2 ivggt on days 1, 8, repeated every 21 days.
  Other Names: Cisplatin
  Arms: Irinotecan plus Cisplatin

SUMMARY:
The aim of this study is to investigate the efficacy, safety, and survival benefit of etoposide plus cisplatin and irinotecan plus cisplatin in first-line therapy of non-primary pancreatic metastatic and/or unresectable gastrointestinal neuroendocrine tumor G3 type. In addition, the investigators will explore the resistance mechanisms of gastrointestinal neuroendocrine tumor G3, and screen out biomarkers that can predict the efficacy of chemotherapy.

DETAILED DESCRIPTION:
The prognosis of gastrointestinal neuroendocrine tumor G3 type patients who cannot be surgically resected is poor. The median overall survival (OS) is only 6-10 months, and the 3-year survival rate is less than 10%. Among the neuroendocrine tumors of the digestive system, only pancreatic neuroendocrine tumor has a standard treatment strategy, and there is a lack of prospective clinical research data on other gastrointestinal neuroendocrine tumors. According to the chemotherapy regimen of small cell lung cancer, etoposide plus cisplatin or irinotecan plus cisplatin is the choice of rescue therapy for advanced non-surgical or metastatic neuroendocrine tumor G3 type. However, prospective studies are needed to confirm whether there are differences in efficacy and safety between the two chemotherapy regimens. The aim of this study is to investigate the efficacy, safety, and survival benefit of etoposide plus cisplatin and irinotecan plus cisplatin in first-line therapy of non-primary pancreatic metastatic and/or unresectable gastrointestinal neuroendocrine tumor G3 type. In addition, the investigators will explore the resistance mechanisms of gastrointestinal neuroendocrine tumor G3, and screen out biomarkers that can predict the efficacy of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18-75 years old, male or female. 2. Confirmed non-primary pancreatic metastatic and/or unresectable gastrointestinal neuroendocrine tumor G3 type patients by histopathological and imaging examinations.

  3. ECOG performance status 0-1. 4. Life expectancy ≥ 12 weeks. 5. A histological specimen can be provided for secondary testing. 6. According to the evaluation criteria of solid tumor efficacy (RESIST 1.1), there should be at least one measurable lesion (empty organs such as esophagus and stomach cannot be taken as the measurable lesion), and the measurable lesion should not have received local treatment such as radiotherapy (the lesion located in the previous radiotherapy area is also selected as the target lesion if the lesion progression is confirmed).

  7. Never received system treatment before, including cytotoxic drugs. For patients who have received adjuvant or neoadjuvant chemotherapy appears recurrence or metastasis more than 6 months from accepting the last dose of chemotherapy drugs can be screened.

  8. The main organ function meets the following criteria within 7 days before treatment:
  1. Blood routine examination criteria (without blood transfusion within 14 days): hemoglobin (HB) ≥ 90g/L, the absolute value of neutrophils (ANC) ≥ 1.5 x 10^9/L, platelet (PLT) ≥ 80 x 10^9/L.
  2. Biochemical examinations must meet the following criteria: total bilirubin (TBIL) ≤ 1.5 x upper limit of normal (ULN), alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 2.5 x ULN, serum creatinine (Cr) ≤ 1.5 x ULN or creatinine clearance (CCR) ≥ 60 mL/min.
  3. Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ normal low limit (50%).

  9. Fertile men and women must use effective contraception during the study period and within 6 months after the end of the study.

  10. Volunteered to participate in the study and signed an informed consent form.

Exclusion Criteria:

* 1.Patients exceeding or currently suffering from other malignant tumors within 5 years, except for cervical cancer in site, non-melanoma skin cancer and superficial bladder tumors (Ta (non-invasive tumor), Tis (in situ carcinoma), and T1 (tumor infiltrating basement membrane)); Patients with rapid progress within 3 months.

  2. History of gastrointestinal perforation and/or fistula within 6 months prior to the first administration.

  3. Patients who had received radiotherapy for tumor target lesions within 4 weeks before enrollment.

  4. History of immunodeficiency disease, including HIV positive and other acquired or congenital immunodeficiency diseases.

  5. Allergic reactions and drug adverse reactions:
  1. A history of allergy to the ingredients of the study drug;
  2. Any contraindication to any study drug (etoposide, irinotecan and cis-platinum) in the chemotherapy regimen.

  6. Significantly malnourished patients. Exclusion is performed if the patient is receiving intravenous fluids or is required to be hospitalized for continuous infusion therapy. Patients with good nutrition control ≥ 28 days can be enrolled before randomization.

  7. Any severe and/or uncontrolled disease, including:
  1. Patients with hypertension whose blood can't be well controlled by antihypertensive drugs (systolic blood pressure ≥ 150 mmHg, diastolic blood pressure ≥ 100 mmHg).
  2. Grade 1 or higher myocardial ischemia or myocardial infarction, arrhythmia (including QTc ≥ 480 ms) or grade 2 and above congestive heart failure according to New York Heart Association (MYHA) classification.
  3. Severe or uncontrolled disease or active infection (≥ CTC AE grade 2), which the investigators believe may increase the risk associated with patient participation and drug administration.
  4. Renal failure requiring hemodialysis or peritoneal dialysis.
  5. Patients of diabetes who have poor glycemic control (fasting blood glucose (FBG) > 10 mmol/L).
  6. Patients of seizures requiring treatment. 8. Patients with gastrointestinal disease such as intestinal obstruction (including incomplete intestinal obstruction) or those who may meet gastrointestinal bleeding, perforation obstruction.

  9. Patients who underwent surgical treatment, incision biopsy or significant traumatic injury within 28 days prior to enrollment.

  10. Any bleeding event ≥ CTC AE grade 3 or unhealed wounds, ulcers or fractures in 4 weeks prior to enrollment.

  11. Arterial/venous thrombosis events within 3 months, such as cerebrovascular accidents (including transient ischemic attacks), deep venous thrombosis and pulmonary embolism.

  12. Patients who prepared or accepted previously allogeneic organ or bone marrow transplantation, including liver transplantation.

  13. Concomitant disease that seriously harms the patient's safety or affects the patient's completion of the study according to the investigator's judgment.

  14. Patients cannot provide histological specimens for secondary test. 15. Patients who have a history of psychotropic substance abuse and are unable to quit or have a mental disorder.

  16. Urine routine showed urinary protein ≥ 2 + and 24-hour urine protein quantitation > 1.0 g.

  17. Patients with brain metastases. 18. Patients who have participated in other anti-tumor drug clinical trials within 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 2 years
  To compare objective response rate of the two arms from date of anti-cancer therapy until progression
Progression-free Survival (PFS) | up to 2 years
  From the first day of treatment until the date of first documented progression or date of death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) | up to 2 years
  From the first day of treatment to death or last survival confirm date
Number of Participants with Treatment-related Adverse Events | up to 2 years
  Treatment-related adverse events will be assessed by CT CAE v4.0
Assessment of Health-related quality of life | up to 2 years
  Quality of Life Questionnaire (QLQ-C30) will be evaluated since treatment begins. At the end of the trail, the differences between the two indicators will be compared with Mixed-effects model repeated measures (MMRM), where the baseline is scored as a covariant and the treatment group as a fixed variable. In addition, the baseline values of the two scores, the value of each visit, and the change value of the baseline will be statistically described.

CONTACTS AND LOCATIONS:
Overall Officials: Baoxia He, Study Director — Henan Cancer Hospital